CLINICAL TRIAL: NCT04747587
Title: Non-use après Accident Vasculaire cérébral : Influence de la Force et de la précision du Geste à Fournir Lors Des Mouvements du Membre supérieur parétique
Brief Title: Non-use After Stroke: Influence of Applied Force and Precision When Reaching With the Paretic Upper Limb
Acronym: OPTISTROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2020-1/JF-01; NCT04747587 (Other: ANSM)
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Non-use; Compensation; Weakness; Optimal control
MeSH Terms: conditions — Stroke; Asthenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with stroke (Experimental)
  Interventions: Other: Reaching Session
- Controls (Experimental)
  Interventions: Other: Reaching Session

INTERVENTIONS:
Other: Reaching Session — Two x 45 minutes sessions of reaching tasks. Patients in the stroke group will perform the task with the paretic arm using a weight reduction system, allowing movement in the horizontal plane.
  Subjects in the control group will perform the task with the randomly selected arm weighted at 80% of their maximum voluntary shoulder torque

SUMMARY:
After a stroke, 80% of patients have an upper limb deficit, limiting activity. Some develop a non-use: they can, but do not, use their paretic limb. Non-use is a general phenomenon applied to all situations where the patient applies unnecessary compensation. Several rehabilitation techniques are effective to counter non-use, but there is insufficient knowledge to choose the most suitable technique. Optimal control theory could help guide these choices. It assumes that the chosen coordination satisfies the constraints of the task (force, amplitude, tolerance) while reducing the cost of the movement. This study will assess non-use by anticipating the sensitivity to the constraints of force and precision deduced from the logic of optimal control. The study authors expect to observe a weakness effect: in a reaching task (i.e. when the person has to touch an object placed in front of them), lightening the paretic arm makes it possible to reduce non-use, and a precision effect: in a reaching task, non-use increases with the required spatial precision.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria specific to the stroke group:

* Patient having had a 1st stroke
* Patient whose stroke occurred more than a month ago.
* Patient having had a supratentorial stroke
* Patient able to touch the opposite knee with the paretic arm

Inclusion criteria specific to the control group:

* Subject who has never had a stroke
* Subject without motor or orthopedic impairment of the upper limbs and in particular of the shoulder

General inclusion criteria:

* Subject who has given free and informed consent.
* Subject who signed the consent form.
* Subject affiliated or beneficiary of a health insurance plan.

Exclusion criteria:

* Pregnant, parturient or breastfeeding subject.
* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient with cognitive disorders incompatible with a good understanding of the use of the device
* Patient with other neurological or osteoarticular history that may limit the performance of the task - criterion left to the deiscretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the modifications of the proximal non-use after stroke on the paretic side according to the extent of force constraint | Inclusion
  Proximal Arm Non Use (PANU) score (%): A significant PANU (> 7.5%) indicates non-use

SECONDARY OUTCOMES:
Evaluate the modifications of the proximal non-use after stroke on the paretic side according to the precision required | Inclusion
  PANU score (%): Physiological non-use considered as a decrease in PANU due to to the increase in the size of the target; A psychological non-use considered as absence of decrease in PANU, regardless of the condition
Evaluate the modifications of the proximal non-use in the control subjects according to the constraints of force or precision | Inclusion
  PANU score (%) of force and precision
Evaluate the level of neuromuscular activation during reaching | Inclusion
  % Voluntary Maximum Contraction (VMC) of anterior and intermediate part of the deltoid, biceps brachii and pectoralis major
Model the constraints and costs explaining non-use patient by patient, to distinguish between physiological and psycho-behavioral non-use | Inclusion
  Weight-over-force ratio of the arm (Ratio between 0 & + ∞)
Time since stroke (acute, subacute or chronic phase) | Inclusion
  months
Intensity of arm deficit | Inclusion
  Fugl-Meyer Upper Extremity score ) (score between 0 and 66)
height of the target | Inclusion
  Evaluate changes in the proximal non-use after stroke on the paretic side according to the height of the target to be reached with PANU score (%) : A significant PANU (> 7.5%) indicates non-use

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Froger, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes

IPD SHARING:
Plan to Share IPD: Yes
Anonymised raw datasets and code used for the analysis will be available on reasonable request.
Supporting Information: Analytic Code